CLINICAL TRIAL: NCT02066246
Title: Investigation of the Possible Advantages of the AirSeal-system Compared to Conventional CO2 Insufflation Systems in Terms of Lung Function and Hemodynamics in Robot-assisted Laparoscopic Radical Prostate Ectomy
Brief Title: Lung Function After Robot-assisted Radical Prostate Ectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Prostate Center North West Department of Urology and Pediatric Urology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ANA-UKE-PV4374
Record Dates: First submitted 2014-01-22; First posted 2014-02-19 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Lung Function
Keywords: laparoscopic robot-assisted surgery; in steep trendelenburg position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olympus UHI-3 (Sham Comparator): patients are treated with the Olympus UHI-3-CO2-insufflation and trocar system
  Interventions: Device: Olympus UHI-3
- AirSeal (Active Comparator): patients are treated with the AirSeal-CO2-insufflator and trocar-system
  Interventions: Device: AirSeal

INTERVENTIONS:
Device: AirSeal — 100 patients are treated with the AirSeal insufflation and trocar system
  Arms: AirSeal
Device: Olympus UHI-3 — 100 patients are treated with a conventional insufflation and trocar system
  Arms: Olympus UHI-3

SUMMARY:
The aim of our study is to investigate if the use of the AirSeal insufflation system impairs the lung function of patients less than a conventional system in patients undergoing robot-assisted laparoscopic radical prostatectomy (RALP). Therefore we examine the lung function before and after surgery.

As a second purpose of the study, in a subgroup, we investigate the influence of the gas insufflators (AirSeal and conventional) on hemodynamics during surgery. Furthermore we study the change in the lung perfusion-ventilation-ratio by using the electric impedance tomography technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for RALP
* Written informed consent
* ≥ 18 years of age

Exclusion Criteria:

* Age under 18 years
* Patients who refuse participating in the study
* Obstructive airway disease (COPD and Asthma)
* Postoperative admission to an intensive or intermediate care unit
* Patients who do not speak German or English

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
forced vital capacity (FVC) | before operation, 1, 24, 120 hours after surgery
forced expiratory volume in one second (FEV1) | before operation, 1, 24, 120 hours after surgery

SECONDARY OUTCOMES:
ventilation parameters | after induction, 30minutes after trendelenburg position, one hour after trendelenburg, two hours after trendelenburg (if operation has not been finished yet), patient in supine position
  peak pressure, positive end-expiratory pressure, end-tidal CO2, respiratory rate are recorded during surgery
hemodynamic parameters | after induction, 30minutes after trendelenburg position, one hour after trendelenburg, two hours after trendelenburg (if operation has not been finished yet), patient in supine position
  global end diastolic volume (GEDV), stoke volume variation (SVV); cardiac index (CI), extravascular lung water index (EVLWI)
electric impedance tomography | after induction, 30minutes after trendelenburg position, one hour after trendelenburg, two hours after trendelenburg (if operation has not been finished yet), patient in supine position

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Reuter, PhD MD, Study Director — Department of Anaesthesiology Center of Anaesthesiology and Intensive Care Medicine University Medical Center Hamburg-Eppendorf University of Hamburg; Alexander März, MD, Principal Investigator — Department of Anaesthesiology Center of Anaesthesiology and Intensive Care Medicine University Medical Center Hamburg-Eppendorf University of Hamburg; Günter Lippert, MD, Principal Investigator — Prostate Cancer Center North West, at St. Antonius-Hospital, Gronau, Germany .; Alexander Haese, PhD MD, Principal Investigator — Martini Clinic, Prostate Cancer Center, University Hospital Hamburg-Eppendorf, Hamburg, Germany.; Jörn Witt, MD, Principal Investigator — Prostate Cancer Center North West, at St. Antonius-Hospital, Gronau, Germany
Locations (2):
- Germany (2):
  - Prostate Cancer Center Northwest, at St. Antonius Hospital Gronau, Gronau
  - Department of Anaesthesiology Center of Anaesthesiology and Intensive Care Medicine University Medical Center Hamburg-Eppendorf University of Hamburg, Hamburg